CLINICAL TRIAL: NCT05655481
Title: Effects of a Home Telerehabilitation Program Via Videoconference in Patients With Pulmonary Arterial Hypertension- Randomized Clinical Trial
Brief Title: Telerehabilitation Program Via Videoconference PAH - Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, LUCIANA MARIA MALOSA SAMPAIO, Professor of the Postgraduate Program in Rehabilitation Sciences, University of Nove de Julho
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAH - Telerehabilitation
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Arterial Hypertension; Cardiovascular Diseases; Respiratory Disease Nursing; Hypertension, Pulmonary; Pulmonary Hypertension
Keywords: Exercise Functional Capacity; Pulmonary Arterial Hypertension; Telerehabilitation; Functional Capacity
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Cardiovascular Diseases; Hypertension, Pulmonary | interventions — Resistance Training; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): AEROBIC TRAINING
  2 training sessions per week for a period of 8 weeks
  Connection platform: WhatsApp
  The research participant will use a 20 cm step on which he will have to go up and down until he reaches the predicted training heart rate.
  Intensity: 60-80% of the maximum heart rate reached at the peak of the incremental step test
  5 minutes warm-up: 60% of maximum heart rate
  20 minutes of Training: 60 to 80% of the maximum heart rate reached at the peak of the incremental step test
  5 minute cool down: 60% of maximum heart rate
  Duration 30 minutes
  RESISTANCE TRAINING
  Devices: Anklet (variable load), these devices will be made available to the research participant
  Exercises for upper limbs, shoulder flexion, elbow flexion and shoulder abduction, and for lower limbs hip flexion and extension.
  Intensity: 70% of the maximum starting load of a 1RM repetition
  3 sets of 8 repetitions
  Duration: 30 minutes
  Interventions: Other: Aerobic and Resistance training with rehabilitation
- Telehealth (Experimental): Guidelines leaflet with health education proposals Explanations about your disease, what it is, psychopathological diagnoses and pharmacological and non-pharmacological treatment), information about the importance of physical activity in your daily life, such as walking, stretching or some daily physical activity according to your preference .
  This group will not receive aerobic or resistance training.
  You will receive telemonitoring twice a week over a period of 8 weeks as a form of teleconsultation in health with the physiotherapist for monitoring throughout the research.
  After this period it will be reassessed.
  Interventions: Other: Health education

INTERVENTIONS:
Other: Aerobic and Resistance training with rehabilitation — Effects of home telerehabilitation program improve functional capacity variables
  Arms: Telerehabilitation
Other: Health education — Telehealth and guidelines for the practice of physical activity and health education
  Arms: Telehealth

SUMMARY:
Pulmonary arterial hypertension (PAH) is a serious, progressive disease that causes pulmonary arterial pressure, significantly affecting functional capacity and quality of life.

Over the last few years, knowledge in pulmonary hypertension has evolved consistently and significantly. New diagnostic and treatment algorithms were combined based on the results of several clinical studies that showed the usefulness of new tools, as well as the effectiveness of new drugs as well as non-pharmacological treatment. The new guidelines felt the benefits of physical exercise in individuals with PAH, with promising results in improving symptoms, exercise capacity, peripheral muscle function and quality of life.

With the COVID 19 pandemic, the complex scenario was for world health, and social distancing made it impossible to carry out individual outpatient rehabilitation, in groups and in person, indicating the need for rehabilitation programs, including physical training, to be adapted to the domicile.

New alternative modes of pulmonary rehabilitation include home-based models and the use of telehealth. Telerehabilitation is the provision of rehabilitation services at a distance, using information and communication technologies. To date, there has been no evaluation of the clinical efficacy or safety of telerehabilitation in the population affected by PAH.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is a type of high blood pressure that affects the arteries in the lungs and the right side of the heart.

In one form of pulmonary hypertension, called PAH, blood vessels in the lungs are narrowed, blocked or destroyed. The damage slows blood flow through the lungs, and blood pressure in the lung arteries rises. The heart must work harder to pump blood through the lungs. The extra effort eventually causes the heart muscle to become weak and fail. In some people, pulmonary hypertension slowly gets worse and can be life-threatening. Although there's no cure for some types of pulmonary hypertension, treatment can help reduce symptoms and improve quality of life.

Several studies show the importance of physical training in patients with PAH. In the study by Meirelles et al. individuals with severe chronic PAH achieved positive results when manifested to physical training, improved the distance walked in the 6-minute walk test (6MWD) by 96±61m after 15 weeks compared to the control group (p<0.001) and several other studies point out the importance of aerobic training for this pulmonary hypertension (PH) population.

However, it is known that exercise limitation in PAH is multifactorial, having right ventricular dysfunction, chronotropic incompetence, ventilatory abnormalities and skeletal muscle dysfunction as causes. mechanical restrictions, poor oxygenation of the skeletal and cerebral muscle, hyperventilation with variations/or increase in the sympathetic impulse.

ELIGIBILITY:
Inclusion Criteria:

* Participants with PAH from group 1 of the HP leaderboard
* Confirmed diagnosis of PAH by cardiac catheterization measurements as defined in group 1, with NHNY functional class I to IV (receiving specific pharmacological therapy for PAH), aged 18 to 70 years
* They are clinically stable without having been hospitalized in the last few weeks.
* Having internet with a data package and knowing how to use WhatsApp to manage telerehabilitation

Exclusion Criteria:

* Requiring continuous oxygen therapy
* Clinical groups 3, 4 and 5
* Significant musculoskeletal disease or limb claudication pain; Psychological or cognitive impairment, psychiatric psychological or mood disorders that may affect your ability to perform the clinical field test
* History of moderate or severe chronic lung disease
* Left heart disease, angina and/or fast heart rate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-04-25 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Change from baseline to 8 weeks
  Oxygen consumption measured during cardiopulmonary testing
6 Minute Walking Test | Change from baseline to 8 weeks
  Distance in meters
Maximum heart rate | Change from baseline to 8 weeks
  Correlate the maximum heart rate of both functional capacity tests
Interchangeable tests | Change from baseline to 8 weeks
  Correlate the distance covered in the six-minute walk test with the number of climbs in the incremental step test

SECONDARY OUTCOMES:
FVC | Change from baseline to 8 weeks
  Lung function - forced vital capacity
FEV1 | Change from baseline to 8 weeks
  Lung function - expiratory volume in 1 second
Health-related quality of life score | Change from baseline to 8 weeks
  scores by EmPHasis-10- health-related quality of life Pulmonary hypertension. Score 0-50

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Malosa Sampaio, Ph.D, Principal Investigator — University of Nove de Julho
Locations (1):
- Luciana Maria Malosa Sampaio, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pandey A, Garg S, Khunger M, Garg S, Kumbhani DJ, Chin KM, Berry JD. Efficacy and Safety of Exercise Training in Chronic Pulmonary Hypertension: Systematic Review and Meta-Analysis. Circ Heart Fail. 2015 Nov;8(6):1032-43. doi: 10.1161/CIRCHEARTFAILURE.115.002130. Epub 2015 Jul 16. PMID 26185169
- [Result] Buys R, Avila A, Cornelissen VA. Exercise training improves physical fitness in patients with pulmonary arterial hypertension: a systematic review and meta-analysis of controlled trials. BMC Pulm Med. 2015 Apr 22;15:40. doi: 10.1186/s12890-015-0031-1. PMID 25896259
- [Result] Ehlken N, Lichtblau M, Klose H, Weidenhammer J, Fischer C, Nechwatal R, Uiker S, Halank M, Olsson K, Seeger W, Gall H, Rosenkranz S, Wilkens H, Mertens D, Seyfarth HJ, Opitz C, Ulrich S, Egenlauf B, Grunig E. Exercise training improves peak oxygen consumption and haemodynamics in patients with severe pulmonary arterial hypertension and inoperable chronic thrombo-embolic pulmonary hypertension: a prospective, randomized, controlled trial. Eur Heart J. 2016 Jan 1;37(1):35-44. doi: 10.1093/eurheartj/ehv337. Epub 2015 Jul 31. PMID 26231884
- [Result] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Pradella CO, Belmonte GM, Maia MN, Delgado CS, Luise AP, Nascimento OA, Gazzotti MR, Jardim JR. Home-Based Pulmonary Rehabilitation for Subjects With COPD: A Randomized Study. Respir Care. 2015 Apr;60(4):526-32. doi: 10.4187/respcare.02994. Epub 2014 Sep 30. PMID 25269680
- [Result] Maron BA, Hess E, Maddox TM, Opotowsky AR, Tedford RJ, Lahm T, Joynt KE, Kass DJ, Stephens T, Stanislawski MA, Swenson ER, Goldstein RH, Leopold JA, Zamanian RT, Elwing JM, Plomondon ME, Grunwald GK, Baron AE, Rumsfeld JS, Choudhary G. Association of Borderline Pulmonary Hypertension With Mortality and Hospitalization in a Large Patient Cohort: Insights From the Veterans Affairs Clinical Assessment, Reporting, and Tracking Program. Circulation. 2016 Mar 29;133(13):1240-8. doi: 10.1161/CIRCULATIONAHA.115.020207. Epub 2016 Feb 12. PMID 26873944
- [Result] Desai SA, Channick RN. Exercise in patients with pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2008 Jan-Feb;28(1):12-6. doi: 10.1097/01.HCR.0000311502.57022.73. PMID 18277824
- [Result] Hansen H, Bieler T, Beyer N, Kallemose T, Wilcke JT, Ostergaard LM, Frost Andeassen H, Martinez G, Lavesen M, Frolich A, Godtfredsen NS. Supervised pulmonary tele-rehabilitation versus pulmonary rehabilitation in severe COPD: a randomised multicentre trial. Thorax. 2020 May;75(5):413-421. doi: 10.1136/thoraxjnl-2019-214246. Epub 2020 Mar 30. PMID 32229541